CLINICAL TRIAL: NCT06277154
Title: A Phase II Study Evaluating the Safety and Efficacy of MASCT-I Combined With Doxorubicin and Ifosfamide for First-line Treatment in Patients With Advanced Soft Tissue Sarcoma
Brief Title: MASCT-I Combined With Doxorubicin and Ifosfamide for First-line Treatment of Advanced Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HRYZ Biotech Co. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASCT-I-2004
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Leiomyosarcoma; Liposarcoma; Synovial Sarcoma; Angiosarcoma; Undifferentiated Pleomorphic Sarcoma; Epithelioid Sarcoma; Malignant Peripheral Nerve Sheath Tumors; Fibrosarcoma; Pleomorphic Rhabdomyosarcoma; Endometrial Stromal Sarcoma; Desmoplastic Small Round Cell Tumor
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Hemangiosarcoma; Histiocytoma, Malignant Fibrous; Sarcoma; Neurofibrosarcoma; Fibrosarcoma; Sarcoma, Endometrial Stromal; Desmoplastic Small Round Cell Tumor | interventions — Doxorubicin; Injections; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASCT-I+ Doxorubicin+ Ifosfamide (Experimental): The final products of MASCT-I technology are dendritic cells (DC) and effector T cells. DC cells injection will be given via subcutaneous injection, and T cells injection will be given via Intravenous (IV) infusion. Doxorubicin and Ifosfamide will be given per protocol.
  Interventions: Biological: MASCT-I; Drug: Doxorubicin; Drug: Ifosfamide
- Doxorubicin+ Ifosfamide (Active Comparator): Doxorubicin and Ifosfamide will be given per protocol.
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide

INTERVENTIONS:
Biological: MASCT-I — The final products of MASCT-I technology are dendritic cells (DC) and effector T cells.
  Arms: MASCT-I+ Doxorubicin+ Ifosfamide
Drug: Doxorubicin — Commercially approved for cancer treatment
  Other Names: Doxorubicin hydrochloride for Injection
Drug: Ifosfamide — Commercially approved for cancer treatment
  Other Names: Ifosfamide for Injection

SUMMARY:
This study will evaluate the safety and efficacy of MASCT-I combined with Doxorubicin and Ifosfamide for first-line treatment in patients with advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label study to evaluate the safety and efficacy of MASCT-I combined with Doxorubicin and Ifosfamide for first-line treatment in patients with metastatic or recurrent unresectable advanced soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years and≤70 years;
2. According to WHO Classification of Tumours, 5th Edition, Volume 3: Soft Tissue and Bone Tumours, histopathologically or cytologically confirmed unresectable locally advanced or metastatic soft tissue sarcomas, including leiomyosarcoma, liposarcoma, synovial sarcoma, angiosarcoma, undifferentiated pleomorphic sarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumors, fibrosarcoma, pleomorphic rhabdomyosarcoma, endometrial stromal sarcoma, desmoplastic small round cell tumor.
3. No previous treatment with systematic chemotherapy or targeted therapy for advanced soft tissue sarcomas or whose disease progressed after 6months of the end of neoadjuvant or adjuvant therapy.
4. At least one measurable and assessable lesion defined by RECIST 1.1;
5. ECOG performance status of 0-1;
6. Estimated life expectancy≥6 months;
7. Pulmonary function is basically normal;
8. Subjects with organ function as defined below (any blood components and growth factors are not allowed within 14 days before apheresis): a) Hemoglobin ≥90g/L; b) Leukocyte≥3.5x10^9/L; c) The absolute neutrophil count (ANC)>1.5x10^9/L; d) Platelet≥100x10^9/L; e) ALT, AST≤2.5 ULN (Upper Limit of Normal), ALT, AST≤5 ULN for liver metastases; f) ALP≤2.5 ULN; g) Serum total bilirubin≤1.5 ULN; Patients with Gilbert's syndromes (persistent or repeated hyperbilirubinemia [mainly unconjugated bilirubin], in the absence of evidence of hemolysis or liver disease), are allowed to enroll with investigator's agreement; h) Serum urea nitrogen or urea and creatinine≤2.5 ULN; i) Serum albumin≥35g/L; j) PT, APTT, INR≤1.5 ULN (without anticoagulation treatment);
9. Obtain the written informed consent of the patient/legal representative;
10. Subjects with potential fertility must agree to use effective contraceptive measure during and within 6 months after the treatment period. HCG test for female with potential fertility must be negative before the study was included.

Exclusion Criteria:

1. Previous treatment with targeted therapy, radiotherapy (radiotherapy to non-target lesions or disease progressed after radiotherapy could be included.) or other antineoplastic drugs such as anlotinib, gemcitabine, within 4 weeks before randomization, or have received Chinese medicine or proprietary Chinese medicine for anti-tumor treatment within 2 weeks before randomization.
2. Highly differentiated liposarcoma, malignant perivascular epithelioid tumor, protuberant cutaneous fibrosarcoma, extraosseous osteosarcoma, solitary fibroma/hemangiopericytoma, acinous soft tissue sarcoma, extraosseous myxoid chondrosarcoma, gastrointestinal stromal tumor, invasive fibroma, renal angiomyolipoma, malignant mesothelioma, clear cell sarcoma, Ewing's sarcoma, etc., which are not suitable for Doxorubicin+ Ifosfamide (AI) treatment.
3. Previous treatment with anthracyclines or anthraquinones and whose cumulative dose exceeds equivalent 200mg/m2 doxorubicin.
4. Previous treatment with MASCT, or have received other cellular immunotherapy or anti-PD-1, anti-PD-L1 antibody therapy in the past 1 year.
5. Use of immunosuppressive agents or systemic or inhaled local hormones (exceeding 10mg/day prednisone or its equivalent) and were still using them within 2 weeks before randomization.
6. Use of immunomodulators and were still using them within 2 weeks before randomization.
7. Allergic to sodium citrate or human albumin.
8. Subjects with uncontrolled pleural effusion and abdominal effusion requiring repeated drainage and with moderate or higher volume of pericardial effusion.
9. Have known active central nervous system (CNS) or meningeal metastases. Subjects with previously treated brain metastases may participate provided they are stable based on the following: 1) any neurologic symptoms have returned to baseline at least 2 weeks before randomization, 2) no requirement for steroids at least 2 weeks before randomization or receiving low-dose of steroids (Not exceeding 10mg/day prednisone or its equivalent).
10. Have any active autoimmune disease or history of autoimmune disease.
11. Subjects with active tuberculosis.
12. Subjects were infected with hepatitis B virus, hepatitis C virus or HIV, or syphilis.
13. Severe cardiovascular disease, such as: (1) complete left bundle branch block or III atrioventricular block; (2) history of myocardial infarction, angioplasty, coronary artery bypass graft; (3) prolonged QT/QTc interval at baseline (male>450ms, female >480ms); (4) LVEF≤50%; (5) heart failure of NYHA class 2 or higher; (6) poorly controlled hypertension (BP≥150/95 mmHg, despite optimal medical treatment); (7) cardiomyopathy or severe arrhythmia and may have impact on the study based on investigator's judgement.
14. Subjects with history of thrombus or experienced a cerebrovascular accident within 6 months before randomization;
15. Other malignant tumors (except cured skin basal cell carcinoma, prostate carcinoma in situ and cervical carcinoma in situ) in the past 5 years;
16. Known history of organ transplantation or ready to receive an organ transplantation;
17. Subjects who have undergone major surgery or traumatic injury within 4 weeks before randomization;
18. Those who have a history of alcohol dependence, psychotropic substance abuse and cannot abstain or have mental disorders.
19. Surgery for soft tissue sarcoma is planned during the study.
20. Subjects have participated in another investigational trial within 4 weeks before randomization.
21. Any condition that the investigator considers to be prejudicial to the subject or to the subject's inability to meet or perform the study requirements exists.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 3 years
  The time from the date of randomization to the first occurrence of radiological progression or death, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  The time from the date of randomization to the date of death from any cause.
Objective Response Rate (ORR) | 3 years
  The percentage of participants with complete response (CR) or partial response (PR) via investigator assessment per RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.1 relative to the total number of participants in the analysis population.
Disease Control Rate (DCR) | 3 years
  The percentage of participants with CR, PR, or stable disease (SD) relative to the total number of participants within the analysis population as determined by Investigators per RECIST v1.1.
Duration of response (DoR) | 3 years
  The time from first documentation of response of PR or better to first documentation of disease progression or death from any cause, whichever comes first.
Adverse events and serious adverse events | 3 years
  All adverse events and serious adverse events during the study
Adverse events and serious adverse events related to MASCT-I | 3 years
  All adverse events and serious adverse events related to MASCT-I during the study
Rate and severity of clinically-significant abnormalities in laboratory testings | 3 years
  Clinically-significant abnormalities in laboratory testings.

OTHER OUTCOMES:
Immune response to tumor-associated antigens | 3 years
  Measured by enzyme linked immunospot assay

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, Principal Investigator — Sun Yat-sen University; Zhang Xing, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No